CLINICAL TRIAL: NCT01013740
Title: A Phase II, Randomised, Multi-Centre Study Evaluating Lapatinib in Combination With Vinorelbine or Capecitabine in Women With ErbB2 Overexpressing Metastatic Breast Cancer
Brief Title: Lapatinib in Combination With Vinorelbine
Acronym: VITAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLAP016A2205 / 112620
Record Dates: First submitted 2009-10-29; First posted 2009-11-16 (Estimated); Results first posted 2013-07-18 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-03

CONDITIONS: Cancer
Keywords: Neoplasms, Breast
MeSH Terms: conditions — Neoplasms; Breast Neoplasms | interventions — Vinorelbine; Lapatinib; Capecitabine

STUDY DESIGN:
Intervention Model Description: After disease progression in the Randomized Phase (in which participants received lapatinib plus vinorelbine), participants were given the option of crossing over to the alternative treatment arm (lapatinib plus capecitabine), and continuing in a post-progression Cross-over Phase.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lapatinib + Vinorelbine (Experimental): Lapatinib + Vinorelbine
  Interventions: Drug: Vinorelbine; Drug: Lapatinib
- Lapatinib + Capecitabine (Active Comparator): Lapatinib + Capecitabine
  Interventions: Drug: Lapatinib; Drug: Capecitabine

INTERVENTIONS:
Drug: Vinorelbine — Vinorelbine
  Arms: Lapatinib + Vinorelbine
Drug: Lapatinib — Lapatinib
Drug: Capecitabine — Capecitabine
  Arms: Lapatinib + Capecitabine

SUMMARY:
This is a randomized, parallel-arm, open-label, multi-centre, Phase II study to determine the efficacy and safety of lapatinib in combination with vinorelbine or capecitabine in women with ErbB2 overexpressing metastatic breast cancer (MBC) who have received no more than one chemotherapeutic regimen in the metastatic setting.

DETAILED DESCRIPTION:
Approximately 105 subjects will be enrolled in the study and randomized 2:1 to one of the following regimens Arm A (n=70): Lapatinib 1250 mg orally once daily continuously plus Vinorelbine 20mg/m2 intravenously (IV) on day 1 and 8, every third week, or Arm B (n=35): Lapatinib 1250 mg orally once daily (QD) continuously plus Capecitabine 2000 mg/m2/day orally in 2 doses 12 hours apart on days 1-14 every third week. Randomization will be stratified according to the following variables: 1) Prior receipt of therapy for metastatic breast cancer (Yes or No), and 2) Site of metastatic disease (Visceral/Soft tissue or Bone-only). Subjects will receive randomized study treatment until disease progression or discontinuation of study treatment due to unacceptable toxicity, withdrawal of consent, lost to follow up, or death. All subjects who discontinue study treatment without documented progression will continue to be followed for progression according to protocol-schedule until new anti-cancer therapy is initiated and/or progression or death is documented. Survival data will be collected for all subjects to ensure a minimum of 18 months survival data. This study will include a safety run-in phase for approximately the first 30 subjects (20 randomized to lapatinib and vinorelbine; 10 to lapatinib and capecitabine).

ELIGIBILITY:
Inclusion Criteria :

* Signed informed consent prior to registration.
* Considered by the investigator to have a life expectancy of ≥12 weeks.
* Subjects must be female and have histologically - confirmed invasive breast cancer with Stage IV disease at primary diagnosis or at relapse after curative - intent surgery.
* Documented overexpression of ErbB2
* Subjects should have progressive disease following prior therapy which may include anthracyclines, taxanes, and trastuzumab.
* Females aged ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 1.
* Subjects must have adequate organ and marrow function
* Subjects must have a cardiac ejection fraction of at least 50% and within the institutional range of normal.
* Radiotherapy prior to initiation of study medication is allowed to a limited area ( e . g . , palliative therapy ) , if it is not the sole site of disease.
* Subjects with stable central nervous system (CNS) metastases are permitted.
* Subject must be free of gastrointestinal diseases or any other conditions that impede swallowing, retaining, and absorption of oral medications.
* Bisphosphonate therapy for bone metastases is allowed; however, treatment must be initiated prior to the first dose of study medication. Prophylactic use of bisphosphonates in subjects without bone disease, except for the treatment of osteoporosis, is not permitted.

Exclusion Criteria:

* Subjects taking prohibited medications are not eligible for the study.
* Therapy with lapatinib, vinorelbine, or capecitabine prior to randomization into this study.
* Prior therapy with more than one chemotherapeutic regimen for metastatic breast cancer.
* Concurrent anticancer or concomitant radiotherapy treatment.
* History of uncontrolled or symptomatic angina; history of arrhythmias requiring medications ; clinically significant myocardial infarction < 6 months from study entry; uncontrolled or symptomatic congestive heart failure; ejection fraction below the institutional normal limit; or any other cardiac condition, which in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient.
* Have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).
* Use of an investigational drug within 30 days or 5 half - lives, whichever is longer, preceding the first dose of investigational treatment, or, concurrent treatment with an investigational agent or participation in another clinical trial involving investigational agents.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to any of the agents used in this study or their excipients that in the opinion of the investigator or GSK Medical Monitor contraindicates their participation.
* Known deficiency for the enzyme dihydropyrimidine dehydrogenase (DPD).
* Known history of uncontrolled inter - current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness / social situations that would limit compliance with study requirements.
* Concurrent disease or condition that would make the subject inappropriate for study participation , or any serious medical disorder that would interfere with the subject's safety.
* Pregnant or lactating females at any time during the study (due to the potential teratogenic or abortifacient effects of lapatinib and breastfeeding).
* Subjects with diseases affecting gastrointestinal function resulting in an inability to take oral medication , including ; malabsorption syndrome, disease significantly affecting gastrointestinal function , or resection of the stomach , small bowel , or colon. Subjects with inflammatory bowel disease or ulcerative colitis are also excluded.
* Peripheral neuropathy of Grade 2 or greater.
* Unresolved or unstable, serious toxicity from prior administration of another investigational drug and / or of prior cancer treatment.
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2009-11-25 (Actual); Primary Completion 2012-08-21 (Actual); Study Completion 2016-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (49):
- Bulgaria (3):
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Chile (2):
  - Novartis Investigative Site, Santiago, RegiÃ³n Metro de Santiago
  - Novartis Investigative Site, ViÃ±a Del Mar, ValparaÃ-so
- France (4):
  - Novartis Investigative Site, Bayonne
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, NÃ®mes Cedex 9
  - Novartis Investigative Site, Saint-Cloud
- Germany (11):
  - Novartis Investigative Site, Rheinfelden, Baden-Wurttemberg
  - Novartis Investigative Site, MÃ¼nchen, Bavaria
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Bad Nauheim, Hesse
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Düsseldorf, North Rhine-Westphalia
  - Novartis Investigative Site, Mönchengladbach, North Rhine-Westphalia
  - Novartis Investigative Site, Velbert, North Rhine-Westphalia
  - Novartis Investigative Site, Mainz, Rhineland-Palatinate
  - Novartis Investigative Site, Chemnitz, Saxony
  - Novartis Investigative Site, Berlin, State of Berlin
- Greece (3):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Heraklion,Crete
  - Novartis Investigative Site, Thessaloniki
- Italy (7):
  - Novartis Investigative Site, Brindisi, Apulia
  - Novartis Investigative Site, Genoa, Liguria
  - Novartis Investigative Site, Brescia, Lombardy
  - Novartis Investigative Site, Turin, Piedmont
  - Novartis Investigative Site, Catania, Sicily
  - Novartis Investigative Site, Ancona, The Marches
  - Novartis Investigative Site, Verona, Veneto
- Mexico (2):
  - Novartis Investigative Site, Monterrey, Nuevo LeÃ³n
  - Novartis Investigative Site, Oaxaca City, Oaxaca
- Poland (7):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Gliwice
  - Novartis Investigative Site, Konin
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Warsaw
- Serbia (2):
  - Novartis Investigative Site, Belgrade
  - Novartis Investigative Site, Kamenitz
- Spain (8):
  - Novartis Investigative Site, Fuenlabrada (Madrid)
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Marbella
  - Novartis Investigative Site, Pamplona
  - Novartis Investigative Site, Reus
  - Novartis Investigative Site, Segovia
  - Novartis Investigative Site, Vigo (Pontevedra)
  - Novartis Investigative Site, Zamora

REFERENCES:
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241
- [Derived] Janni W, Sarosiek T, Karaszewska B, Pikiel J, Staroslawska E, Potemski P, Salat C, Brain E, Caglevic C, Briggs K, Mahood K, DeSilvio M, Marini L, Papadimitriou C. Final overall survival analysis of a phase II trial evaluating vinorelbine and lapatinib in women with ErbB2 overexpressing metastatic breast cancer. Breast. 2015 Dec;24(6):769-73. doi: 10.1016/j.breast.2015.08.005. Epub 2015 Sep 16. PMID 26384789

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the Randomized Phase (RP), participants were treated until disease progression (PD) or discontinuation of treatment due to unacceptable toxicity, withdrawal of consent, lost to follow-up, or death. After PD in the RP, participants were given the option of crossing over to the alternative treatment arm in a post-progression Cross-over Phase (CP).
Groups:
- Lapatinib + Capecitabine in RP; Lapatinib + Vinorelbine in CP: Participants received a daily dose of 5 tablets of lapatinib (1250 milligrams [mg]) continuously at approximately the same time every day, either 1 hour (or more) before food or 1 hour (or more) after food. Participants also received capecitabine 2000 mg per meters squared (mg/m^2) per day, divided and administered orally twice daily, 12 hours apart, for 14 days, every 21 days. Capecitabine was taken with food or within 30 minutes after food with approximately 200 milliliters (mL) of water. After disease progression in the Randomized Phase (in which participants received lapatinib plus vinorelbine), participants were given the option of crossing over to the alternative treatment arm (lapatinib plus capecitabine), and continuing in a post-progression Cross-over Phase.
- Lapatinib + Vinorelbine in RP; Lapatinib + Capecitabine in CP: Participants received a daily dose of 5 tablets of lapatinib (1250 mg) at approximately the same time every day, either 1 hour (or more) before food or 1 hour (or more) after food. Participants also received an intravenous (IV) infusion of vinorelbine 20 mg/m^2 over the course of 5 to 10 minutes on Days 1 and 8 of a 21-day treatment cycle. After disease progression in the Randomized Phase (in which participants received lapatinib plus capecitabine), participants were given the option of crossing over to the alternative treatment arm (lapatinib plus vinorelbine), and continuing in a post-progression Cross-over Phase.
Period: Overall Study
Arm/Group | Lapatinib + Capecitabine in RP; Lapatinib + Vinorelbine in CP | Lapatinib + Vinorelbine in RP; Lapatinib + Capecitabine in CP
Started | 37 (13 participants (par.) experiencing PD in the RP elected to enroll in the optional CP.) | 75 (29 participants experiencing PD in the RP elected to enroll in the optional CP.)
Ongoing | 0 | 0
Completed | 26 (Completion also = 18 mos.of a new anti-cancer therapy initiation +/or progression of disease) | 56 (Completion also = 18 mos.of a new anti-cancer therapy initiation +/or progression of disease)
Not Completed | 11 | 19
Not completed — Lost to Follow-up | 3 | 5
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 2 | 10
Not completed — study close / terminated : done in error | 2 | 1
Not completed — Missing | 2 | 1
Not completed — Ongoing: Study records not completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lapatinib + Capecitabine in RP; Lapatinib + Vinorelbine in CP | Lapatinib + Vinorelbine in RP; Lapatinib + Capecitabine in CP | Total
Number analyzed (Participants) | 37 | 75 | 112
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.5 (10.90) | 57.7 (10.23) | 57.6 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 75 | 112
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 36 | 74 | 110
  Native Hawaiian or other Pacific Islander & White | 1 | 0 | 1
  African American/African Heritage | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) in the Randomized Phase
Description: PFS is defined as the time from randomization until the earliest date of disease progression (PD) or death due to any cause, if sooner. PD is defined as at least a 20 % increase in the sum of the longest diameter (LD) of target lesions, taking as a reference the smallest sum LD recorded since the treatment started or the appearance of >=1 new lesion.
Time Frame: From randomization until disease progression, death, or discontinuation from the study (average of 27 study weeks)
Population: ITT Population: participants who were randomized to study treatment, regardless of whether they actually received study medication
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Lapatinib Plus Capecitabine: Participants received a daily dose of 5 tablets of lapatinib (1250 milligrams [mg]) continuously at approximately the same time every day, either 1 hour (or more) before food or 1 hour (or more) after food. Participants also received capecitabine 2000 mg per meters squared (mg/m^2) per day, divided and administered orally twice daily, 12 hours apart, for 14 days, every 21 days. Capecitabine was taken with food or within 30 minutes after food with approximately 200 milliliters (mL) of water.
- Lapatinib Plus Vinorelbine: Participants received a daily dose of 5 tablets of lapatinib (1250 mg) at approximately the same time every day, either 1 hour (or more) before food or 1 hour (or more) after food. Participants also received an intravenous (IV) infusion of vinorelbine 20 mg/m^2 over the course of 5 to 10 minutes on Days 1 and 8 of a 21-day treatment cycle.
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Vinorelbine
Number analyzed (Participants) | 37 | 75
months | 6.2 [4.4 to 8.3] | 6.2 [4.2 to 8.8]
Statistical Analysis 1: Comparison: Lapatinib Plus Capecitabine vs Lapatinib Plus Vinorelbine; Test type: Superiority or Other; Hazard Ratio (HR) = 0.84, 95% CI [0.53 to 1.35] — The Pike estimator of the treatment HR was based on the log rank test

2. Secondary Outcome: Number of Participants With Overall Response (OR), as Assessed by the Investigator in the Randomized Phase
Description: OR is defined as the number of participants achieving either a confirmed complete response (CR: the disappearance of all target lesions [TLs]) or partial response (PR: a >=30% decrease in the sum of the longest diameter [LD] of the TLs, taking as reference the baseline sum LD) as assessed by the investigator as the best OR.
Time Frame: From randomization until disease progression, death, or discontinuation from the study (average of 27 study weeks)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Vinorelbine
Number analyzed (Participants) | 37 | 75
participants | 13 | 15

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to the date of death due to any cause. Participants who had not died were censored at the date of the last adequate tumor assessment at the time of the cut-off.
Time Frame: From the date of randomization until death (average of 55 study weeks)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Vinorelbine
Number analyzed (Participants) | 37 | 75
months | 19.4 [16.4 to 27.2] | 24.3 [16.4 to NA] — The upper limit of the 95% confidence interval (CI) could not be determined (not reached) because there were not enough events to be able to calculate the upper limit of the CI.

4. Secondary Outcome: Duration of Response (DOR) in the Randomized Phase
Description: DOR is defined as the time from the first documented evidence of response (CR or PR) until the first documented sign of disease progression (a >=20% increase in the sum of the LD of TLs, taking as reference the smallest sum LD recorded since the treatment started or the appearance of >=1 new lesion) or death, if sooner. CR=the disappearance of all TLs. PR=a >=30% decrease in the sum of the LD of target lesions, taking as a reference the Baseline sum LD.
Time Frame: From the time of the first documented confirmed complete or partial response until disease progression or death, if sooner (average of 27 study weeks)
Population: ITT Population. Only participants with a confirmed CR or PR were assessed for duration of response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Vinorelbine
Number analyzed (Participants) | 13 | 15
months | 10.8 [4.3 to NA] — The upper limit of the 95% confidence interval (CI) could not be determined (not reached) because there were not enough events to be able to calculate the upper limit of the CI. | 6.7 [4.6 to 8.3]

5. Secondary Outcome: Time to Response in the Randomized Phase
Description: Time to response is defined as the time from randomization until the first documented evidence of CR (the disappearance of all TLs) or PR (a >=30% decrease in the sum of the LD of the TLs, taking as a reference the basline sum LD) (whichever status is recorded first). When tumor response was confirmed at a repeat assessment, the time to response was taken to be the first time that the response was observed.
Time Frame: From randomization until the time of the first documented confirmed CR or PR (average of 27 study weeks)
Population: ITT Population. Only participants with a confirmed CR or PR were assessed for time to response.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Vinorelbine
Number analyzed (Participants) | 13 | 15
weeks | 9.3 [9.1 to 10.0] | 9.4 [9.0 to 10.1]

6. Secondary Outcome: Number of Participants With Clinical Benefit (CB) in the Randomized Phase
Description: CB is defined as the the number of participants achieving either a confirmed CR or PR or having stable disease (SD) for at least 24 weeks (i.e., approximately 6 months). CR=the disappearance of all TLs. PR=a >=30% decrease in the sum of the LD of TLs, taking as a reference the Baseline sum LD. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD=at least a 20% increase in the sum of the LD of target lesions, taking as a reference the smallest sum LD recorded since the treatment started or the appearance of >=1 new lesion). Participants with unknown or missing responses were treated as non-responders.
Time Frame: From randomization until disease progression, death, or discontinuation from the study (average of 27 study weeks)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Vinorelbine
Number analyzed (Participants) | 37 | 75
participants | 18 | 29
Statistical Analysis 1: Comparison: Lapatinib Plus Capecitabine vs Lapatinib Plus Vinorelbine; Test type: Superiority or Other; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.63 to 3.58]

7. Secondary Outcome: Area Under the Concentration-time Curve Over the Dosing Interval (AUC-tau) for Vinorelbine
Description: AUC-tau is defined as the area under the concentration-time curve over a dosing interval at steady state, where tau is the length of the dosing interval. The AUC is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption. Pharmacokinetic (PK) parameters were to be assessed in an optional sub-study. No participants were enrolled in this optional sub-study; thus, no PK data are available.
Time Frame: Days 1 and 8; 0 to 24 hours post-dose
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Vinorelbine
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Maximum Concentration (Cmax) for Vinorelbine
Description: Cmax is defined as the maximum observed plasma or serum concentration after administration of the drug. PK parameters were to be assessed in an optional sub-study. No participants were enrolled in this optional sub-study; thus, no PK data are available.
Time Frame: Days 1 and 8; 0 to 24 hours post-dose
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Vinorelbine
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants With Grade 4 and Grade 5 Adverse Events (AE)
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Grades: 0 = no AE or within normal limits; 1 = mild AE; 2 = moderate AE; 3 = severe and undesirable AE; 4 = life-threatening or disabling AE; 5 = death related to AE.
Time Frame: From randomization until disease progression, death, or discontinuation from the study (average of 55 study weeks)
Population: Safety Population: participants who received at least one dose of study medication, based on the actual treatment received
Measure: Number; unit: participants
Arm/Group | Lapatinib Plus Capecitabine | Lapatinib Plus Vinorelbine
Number analyzed (Participants) | 37 | 75
participants
  Helicobacter gastritis, Grade 4 | 1 | 0
  Neutropenia, Grade 4 | 0 | 9
  Leukopenia, Grade 4 | 0 | 1
  Febrile neutropenia, Grade 4 | 0 | 1
  Mucosal inflammation, Grade 4 | 0 | 1
  Pulmonary embolism, Grade 4 | 0 | 1
  Intestinal obstruction, Grade 5 | 0 | 1

ADVERSE EVENTS:
Time Frame: Serious Adverse Events are monitored from date of First Subject First Visit (FSFV) until Last Subject Last Visit (LSLV). All other adverse events are monitored from First Subject First Treatment until LSLV. Initiation Date: 25 November 2009- Completion Date: 21 August 2012
Groups:
- Randomized Phase Lapatinib 1250mg QD + Capecitabine 2000mg/m2: Randomized phase Lapatinib 1250mg QD + Capecitabine 2000mg/m2
- Randomized Phase Lapatinib 1250mg QD + Vinorelbine 20mg/m2: Randomized phase Lapatinib 1250mg QD + Vinorelbine 20mg/m2
- Crossover Phase Lapatinib 1250mg QD + Capecitabine 2000mg/m2: Crossover phase Lapatinib 1250mg QD + Capecitabine 2000mg/m2
- Crossover Phase Lapatinib 1250mg QD + Vinorelbine 20mg/m2: Crossover phase Lapatinib 1250mg QD + Vinorelbine 20mg/m2
Arm/Group | Randomized Phase Lapatinib 1250mg QD + Capecitabine 2000mg/m2 | Randomized Phase Lapatinib 1250mg QD + Vinorelbine 20mg/m2 | Crossover Phase Lapatinib 1250mg QD + Capecitabine 2000mg/m2 | Crossover Phase Lapatinib 1250mg QD + Vinorelbine 20mg/m2
Serious Adverse Events (participants affected / at risk) | 4/37 | 25/75 | 3/37 | 4/17
Other Adverse Events (participants affected / at risk) | 32/37 | 72/75 | 27/37 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Phase Lapatinib 1250mg QD + Capecitabine 2000mg/m2 (N=37) | Randomized Phase Lapatinib 1250mg QD + Vinorelbine 20mg/m2 (N=75) | Crossover Phase Lapatinib 1250mg QD + Capecitabine 2000mg/m2 (N=37) | Crossover Phase Lapatinib 1250mg QD + Vinorelbine 20mg/m2 (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 10 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Device leakage (Product Issues) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Phase Lapatinib 1250mg QD + Capecitabine 2000mg/m2 (N=37) | Randomized Phase Lapatinib 1250mg QD + Vinorelbine 20mg/m2 (N=75) | Crossover Phase Lapatinib 1250mg QD + Capecitabine 2000mg/m2 (N=37) | Crossover Phase Lapatinib 1250mg QD + Vinorelbine 20mg/m2 (N=17)
Anaemia (Blood and lymphatic system disorders) | 2 | 13 | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 3 | 11 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 3 | 34 | 2 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 2 | 1
Tachycardia (Cardiac disorders) | 2 | 1 | 0 | 0
Ophthalmoplegia (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 7 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 6 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 6 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 21 | 35 | 7 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 6 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 20 | 6 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 4 | 13 | 0 | 0
Asthenia (General disorders) | 5 | 10 | 3 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 17 | 1 | 2
Inflammation (General disorders) | 0 | 1 | 0 | 1
Influenza like illness (General disorders) | 0 | 2 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 9 | 1 | 0
Oedema peripheral (General disorders) | 1 | 7 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 10 | 2 | 2
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 6 | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 4 | 0 | 1
Cystitis (Infections and infestations) | 1 | 2 | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 4 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 5 | 2 | 2 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 5 | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 8 | 4 | 2
Aspartate aminotransferase increased (Investigations) | 4 | 8 | 5 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 4 | 3 | 1
Blood bilirubin increased (Investigations) | 4 | 0 | 1 | 1
Blood calcium increased (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 5 | 0 | 0
Weight decreased (Investigations) | 2 | 4 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 12 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 9 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 7 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 7 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 8 | 4 | 2
Dizziness (Nervous system disorders) | 0 | 5 | 2 | 0
Headache (Nervous system disorders) | 2 | 8 | 2 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 5 | 2 | 0
Paraesthesia (Nervous system disorders) | 2 | 2 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 8 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 4 | 0 | 1
Vaginal inflammation (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 9 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 6 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 4 | 2 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 24 | 6 | 18 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 15 | 2 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0
Hot flush (Vascular disorders) | 0 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.